CLINICAL TRIAL: NCT05670821
Title: Post-marketing Surveillance of Spesolimab I.V. Infusion in Improvement of Generalized Pustular Psoriasis (GPP) With Acute Symptoms in Japan
Brief Title: PMS of Spesolimab I.V. in GPP Patients With Acute Symptoms
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1368-0093
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with generalized pustular psoriasis (GPP)
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Spesolimab

SUMMARY:
Non-interventional cohort study in patients with newly initiated Spesolimab to evaluate the incidence of adverse drug reactions and to understand generalized pustular psoriasis (GPP) disease activities in the real world setting.

ELIGIBILITY:
Inclusion Criteria:

* GPP patients with acute symptoms who are administered Spesolimab Intravenous (I.V.) Infusion in Japan
* Patients who have never been treated with Spesolimab I.V. Infusion before enrolment

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with generalized pustular psoriasis (GPP).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) | Up to 36 weeks
  Incidence of adverse drug reactions (ADRs). An ADR is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility. Adverse reactions may arise from use of the product within or outside the terms of the marketing authorization or from occupational exposure. Conditions of use outside the marketing authorization include off-label use, overdose, misuse, abuse and medication errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com